# Statistical analysis plan and sample size calculation

## **Official Title:**

The Effect of Chronic Nitrate Supplementation on Acute Mountain Sickness and Exercise Performance in Hypoxia

## **NCT** number

NCT03101904

## **Document Date**

15/10/2015

#### High-altitude headache

RM ANOVA 2x4 RM ANOVA = Total of 8 repeated measures

| | Av correlation | | Meaningful | Effect size | | Sample |
|---|---|---|---|---|---|---|
| | Calculated | Table | difference | Calculated | Table | size |
| Нурохіа | 0.6 | Strong = 0.5 | 14 | 0.7 | Large = 0.57 | 14 |
| | | | 10 | 0.5 | Medium = 0.35 | 23 |
| All data | 0.2 | Weak = 0.3 | 14 | 0.7 | Large = 0.49 | 16 |
| | | | 10 | 0.5 | Large = 0.49 | 16 |
| 4 measures | 0.4 | Weak = 0.3 | 10 | 0.7 | Large = 0.49 | 16 |

#### Calculations (4 measures)

#### **Average correlation**

| | | | Normoxic | | |
|----------|-----|-----|----------|-----|------|
| | | 4 h | 6 h | 8 h | 8 h |
| | 4 h | 1 | 0.4 | 0.4 | |
| Hypoxic | 6 h | | 1 | 0.9 | |
| | 8 h | | | 1 | -0.3 |
| Normoxic | 8 h | | | | 1 |

Average correlation = 0.4

### **Effect size**

Meaningful difference = 10 SD of difference (4-6 h in hypoxia) = 18 Cohen's D = 0.55 Conversion to RM ANOVA effect size = 0.55/(SQRT(1-0.4)) = 0.7 (Stevens, 2002)

A sample size estimation for this analysis indicated that 16 participants were needed to produce an 80% chance of obtaining statistical significance at the 0.05 level (5), based on a minimum important difference of 10 mm (2), a standard deviation of the difference of 18 mm, and an estimated average correlation of 0.4 (data from (3)).

#### Time to exhaustion

t tests - Means: Difference between two dependent means (matched pairs)

Analysis: A priori: Compute required sample size
Input: Tail(s) = Tw

Effect size dz = 0.9090909  $\alpha$  err prob = 0.05Power (1- $\beta$  err prob) = 0.8

Output: Noncentrality parameter  $\delta = 3.1491833$ 

Critical t = 2.2009852

Df = 11 Total sample size = 12

Actual power = 0.8174086

The effect of nitrate supplementation on maximal exercise performance (TTE) was determined by paired samples t-test. A sample size estimation for this analysis indicated that 12 participants were needed to produce an 80% chance of obtaining statistical significance at the 0.05 level for a two-tailed design (1), based on a minimum important difference of 30 seconds and a standard deviation of the difference of 33 seconds (data from (4)). Given the smaller required sample size for this analysis, only 15 participants completed the TTE component of the study.

#### References

- 1. **Bland M**. *Determination of sample size*. 4th ed. Oxford: Oxford University Press, 2015.
- 2. **Kelly AM**. The minimum clinically significant difference in visual analogue scale pain score does not differ with severity of pain. *Emerg Med J* 18: 205–207, 2001.
- 3. **Lawley JS, Oliver SJ, Mullins PG, Macdonald JH**. Investigation of whole-brain white matter identifies altered water mobility in the pathogenesis of high-altitude headache. *J Cereb Blood Flow Metab* 33: 1286–1294, 2013.
- 4. Masschelein E, Van Thienen R, Wang X, Van Schepdael a., Thomis M, Hespel P. Dietary nitrate improves muscle but not cerebral oxygenation status during exercise in hypoxia. *J Appl Physiol* 113: 736–745, 2012.
- 5. **Stevens J**. *Applied multivariate statistics for the social sciences*. 4th ed. New Jersey: Lawrence Erlbaum Associates Inc., 2002.